CLINICAL TRIAL: NCT02416141
Title: Fast-release Orodispersible Tramadol as Analgesia in Termination of Pregnancy by Vacuum Aspiration.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHUTIV2015MDB001
Record Dates: First submitted 2015-03-31; First posted 2015-04-14 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-03

CONDITIONS: Fertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fast release oro-dispersible tramadol (Active Comparator): This group receives a fast release oro-dispersible tramadol 30 minutes before the vacuum aspiration procedure. A paracervical block with a 27-gauge spinal needle with lidocaine will be injected at the the start of the procedure.
  Intervention: use of fast release oro dispersible tramadol 50 mg
  Interventions: Drug: fast release oro dispersible tramadol 50 mg
- Placebo-controlled arm (Placebo Comparator): This group receives a placebo 30 minutes before the vacuum aspiration procedure. A paracervical block with a 27-gauge spinal needle with lidocaine will be injected at the the start of the procedure.
  Intervention: use of placebo

INTERVENTIONS:
Drug: fast release oro dispersible tramadol 50 mg — idem arm 1
  Arms: Fast release oro-dispersible tramadol

SUMMARY:
If a termination of pregnancy procedure is performed by vacuum aspiration our patients receive a paracervical block. Nevertheless these patients are not free of pain. We randomised our patients: one group will receive additional orodispersible tramadol, the other group will receive a placebo.

DETAILED DESCRIPTION:
Patients were administered either 50 mg of fast-release orodispersible tramadol (Meda Pharma, Brussels, Belgium) or placebo 30 min before the procedure. Both, patient and gynecologist were blinded.

Patients underwent the following procedure: a sterile bivalve speculum was introduced into the vagina, then cervix and vagina were washed with an antiseptic solution. The cervix was grasped with a tenaculum and straigthened. A paracervical block was achieved using a 27-gauge spinal needle. Lidocaine was injected and distributed equally around the cervicovaginal junction at 1, 5, 7 and 11 o'clock. The suction curettage was accomplished through the following steps: the cervix was dilated, in function of the gestation, to Hagar number 5 to 11 (Aesculap, Ag and Co. KG, Tuttlingen, Germany); The uterine depth was measured using a hysterometry; suction curettage was performed by using plastic canula (Luneau Sas, France) and a classic suction pump (AMEDA Egnell SA, Switserland). The patients were observed for 2 hours after the curettage procedure.

Patients were asked to rate the pain during different steps of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* - Patients above 18 ans.
* Non desired pregnancy.
* Non evolutive pregnancy.
* Pregnancy < or = 14 weeks of amenorrhea.

Exclusion Criteria:

* - Interruption of pregnancy due to medical reasons
* Patient already included in this study
* Intolerance for Tradonal Odis 50mg

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Will fast-release orodispersible tramadol reduce the pain (VAS) significantly in a vacuum aspiration procedure in this placebo-controlled trial. | 6 to 8 month to include all patients

CONTACTS AND LOCATIONS:
Overall Officials: Michael De Brucker, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UniversitairZB, Jette, Belgium